CLINICAL TRIAL: NCT01297075
Title: Outreach Visits to Optimize Chronic Care Management in General Practice: A Cluster Randomized Trial
Acronym: Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Unit Of General Practice, Copenhagen (Other)
Collaborators: Region Capital Denmark (Other)
Responsible Party: Principal Investigator, Frans Boch Waldorff, Research Associate professor, Research Unit Of General Practice, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: GP00990002
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Disease
Keywords: Health Services Research; Chronic Care; Outreach Visits; Primary care; chronic disease management
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outreach visits (Experimental): Practices allocated to outreach visits may receive up to three outreach visits in order to motivate and support general practice clinics in implementing two chronic care programmes for chronic obstructive Pulmonary disease and Type 2 diabetes.
  Interventions: Behavioral: Outreach visits
- Control (late intervention) (No Intervention): These practices are allocated to outreach visits after the initial evaluation stops at 12 months.

INTERVENTIONS:
Behavioral: Outreach visits — The 16 facilitators in the project attend an educational programme designed to provide them with the necessary skills and tools for the task. The facilitators visit general practice clinics from March 2011 until the end of 2012. Each clinic is offered three visits. The facilitator is to act as a change agent who motivates and helps the clinic team in the process of defining common goals, and choosing the appropriate means for achieving them.
  Arms: Outreach visits

SUMMARY:
The aim of this project is to motivate and support general practice clinics in implementing the visions and recommendations presented in two of the disease specific programmes for chronic care management (for chronic obstructive lung disease and Type 2 diabetes). These programmes describe evidence based treatment and division of tasks between the municipalities, the hospitals and general practice.

The Facilitator Project is funded by The Danish Ministry of Interior and Health.

DETAILED DESCRIPTION:
In a cluster randomized trial the investigators will explore the efficacy of up to three outreach visits by specially trained GPs. Efficacy data are obtained by means of questionnaires at regional databases.

ELIGIBILITY:
Inclusion Criteria:

General Practices working in the capital region in Denmark

Exclusion Criteria:

General Practices where the facilitator works.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 12 month in Annual systematic chronic disease follow up consultations | Month 4, 3, 2 before baseline and month 13,14,15 after baseline (after intervention)
  Change in annual systematic chronic disease controls per person affiliated with a primary care at a period at baseline and at 12 month.

SECONDARY OUTCOMES:
ICPC diagnosis coding | 12 months
  Self reports regarding the use of ICPC diagnosis coding for Type 2 Diabetes and Chronic Obstructive Pulmonary Disease.
Sentinel Data Capture | 12 months
  Application for the electronic Sentinel Data Capture module for overview of patients with chronic diseases.
Stratification | 12 months
  The self reported use of stratification as part of primary care management of patients with chronic diseases
Change from baseline and at 12 month in practices with low performance on annual systematic chronic disease follow up consultations. | Month 4, 3, 2 before baseline and month 13,14,15 after baseline (after intervention)
  Reduction in the number of practices with less than 1% annual systematic chronic disease follow up consultations.

CONTACTS AND LOCATIONS:
Overall Officials: Frans B Waldorff, PhD, Principal Investigator — Research Unit of General Practice
Locations (2):
- Denmark (2):
  - Frans Boch Waldorff, Copenhagen, Capital Area
  - Research Unit of General Practice, Copenhagen, Capital

REFERENCES:
- [Derived] Due TD, Thorsen T, Kousgaard MB, Siersma VD, Waldorff FB. The effectiveness of a semi-tailored facilitator-based intervention to optimise chronic care management in general practice: a stepped-wedge randomised controlled trial. BMC Fam Pract. 2014 Apr 9;15:65. doi: 10.1186/1471-2296-15-65. PMID 24716545